CLINICAL TRIAL: NCT03742076
Title: Effect of Gum Arabic on Gastrointestinal Transit and Permeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18-001008
Record Dates: First submitted 2018-11-05; First posted 2018-11-15 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Prebiotics; Gum Arabic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose prebiotic (Active Comparator): 10 gm gum arabic (powder) with 2 gm fiber powder daily for at least 6 weeks
  Interventions: Dietary Supplement: High-dose prebiotic
- Low-dose prebiotic (Active Comparator): 5 gm gum arabic (powder) with 2 gm fiber powder daily for at least 6 weeks
  Interventions: Dietary Supplement: Low-dose prebiotic
- Placebo (Placebo Comparator): 2 gm powdered fiber daily for at least 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High-dose prebiotic — This is a spray-dried powder, yellowish-white in color, that is dissolvable.
  Other Names: Acacia, gum acacia, acacia gum, gum arabic, arabic gum
  Arms: High-dose prebiotic
Dietary Supplement: Low-dose prebiotic — This is a spray-dried powder, yellowish-white in color, that is dissolvable.
  Other Names: Acacia, gum acacia, acacia gum, gum arabic, arabic gum
  Arms: Low-dose prebiotic
Dietary Supplement: Placebo — Powder fiber supplement, yellowish-white in color, that is dissolvable.
  Other Names: Dextrin fiber powder
  Arms: Placebo

SUMMARY:
The study aims to determine the effect of gum arabic on gut bacteria and GI function.

DETAILED DESCRIPTION:
To compare the effect of placebo, low-dose prebiotic, or high-dose prebiotic on gut microbiota composition and function, GI transit and permeability, and assess development of symptoms or a change in pre-existing symptoms present, in patients with recent history of clinically diagnosed diverticulitis which has been successfully treated.

ELIGIBILITY:
Inclusion Criteria:

1. Recent diagnosis of diverticulitis (within 24 months) and at least 4 weeks post antibiotic use
2. Age 18-80

Exclusion Criteria:

1. Prior history of gastrointestinal surgeries (except appendectomy and cholecystectomy)
2. Known diagnosis of inflammatory bowel disease (Crohn's or ulcerative colitis), microscopic colitis, celiac disease, or other inflammatory condition other than diverticulitis
3. Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
4. Use of NSAIDs or aspirin within the week prior to Visit 2 and Visit 5 (permeability and transit testing visit since NSAIDs affect intestinal permeability)
5. Use of osmotic laxatives one week prior to Visit 2 and for the duration of the study
6. Use of oral corticosteroids within the previous 6 weeks and for the duration of the study
7. Ingestion of artificial sweeteners such as Splenda™ (sucralose), Nutrasweet™ (aspartame), sorbitol, xylitol, lactulose, or mannitol 2 days before and during the permeability testing days, e.g. foods to be avoided are sugarless gums or mints and diet beverages
8. Antibiotic use within 4 weeks of completion of the initial stool kit and/or Visit 2 testing appointment and for the remainder of the study (they can complete the stool kit and Visit 2 after a 4-week washout period)
9. Bowel preparation for colonoscopy less than one week prior to the completion of the first stool kit and Visit 2 and during the remainder of the study
10. Pregnancy or plan to become pregnant within the study timeframe
11. Vulnerable adults
12. Egg allergy or resistant to ingesting eggs
13. Diagnosis of diabetes
14. Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Colonic Transit time | Change is being assessed between baseline and 6 weeks
  The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool. Units: units on a scale

SECONDARY OUTCOMES:
Intestinal Permeability | Change is being assessed between baseline and 6 weeks
  To determine intestinal permeability, urine will be collected for 24 hours after drinking a sugar solution. The 0- to 2-hour urine most closely reflects small intestinal permeability and the 8- to 24-hour urine reflects colonic permeability. HPLC-tandem mass spectrometry will be used for detection of the sugars.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C Kashyap, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials